CLINICAL TRIAL: NCT00189319
Title: Impact of Oral Controlled Release Flecainide Acetate Capsules on Health-Related QoL in Patients With Paroxysmal Atrial Fibrillation
Brief Title: To Evaluate the Impact of Oral Flecainide on Quality of Life in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1478-FLEC
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2006-09

CONDITIONS: Atrial Fibrillation
Keywords: Tambocor; Paroxysmal Atrial Fibrillation; Quality of Life
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Drug: Flecainide controlled release

SUMMARY:
The purpose of this study is to evaluate the management of paroxysmal atrial fibrillation with controlled release flecainide on patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* In sinus rhythm at treatment initiation
* Experienced symptomatic AF episodes
* Left ventricular ejection fraction of at least 40%
* Females of child bearing potential must be using reliable method of contraception

Exclusion Criteria:

* Intolerance and/or failure of previous therapy with flecainide immediate release
* Currently receiving >200mg/day flecainide immediate release
* Severe symptoms during episodes of arrhythmia
* History of other cardiac conditions/abnormalities
* Heart surgery within the last 2 months
* Renal failure
* Pregnant or lactating females
* Significant extra cardiac or systemic disease
* Abnormal electrolyte levels
* Receiving defined cardiac and/or other treatments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-09

PRIMARY OUTCOMES:
To assess the effect of Flecainide CR on patient-perceived health-related QoL (Quality of Life).

SECONDARY OUTCOMES:
assessment of treatment success based on an efficacy/safety composite criterion;
assessment of the relationship between QoL changes and outcomes related to safety and efficacy;
assessment of cardiac safety of Flecainide CR through clinical examination, cardiac adverse events,12-lead paper ECG, and cardiac ultrasonography;
assessment of the non-cardiac safety of Flecainide CR through questioning, non-cardiac adverse events and clinical examination;
evaluation of the course of the disease by the time to the first recurrence of a PAF episode and the subjective symptomatology (duration and severity of PAF episodes).

CONTACTS AND LOCATIONS:
Overall Officials: Salem Kacet, Principal Investigator — Hopital Cardiologique, CHR de Lille, France
Locations (1):
- Hopital Cardiologique, Service de Cardiologique CHR de Lille, Lille, France